CLINICAL TRIAL: NCT00891280
Title: A Phase 1, Multi-Center, Open-Label, Dose-Escalation, Safety, Pharmacokinetic, and Pharmacodynamic Study of CX-4945 Administered Orally to Patients With Advanced Solid Tumors, Castleman's Disease or Multiple Myeloma
Brief Title: Dose-escalation Study of Oral CX-4945
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cylene Pharmaceuticals (Industry)
Responsible Party: Study Director, Cylene Pharmaceuticals Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C4-08-001
Record Dates: First submitted 2009-04-29; First posted 2009-05-01 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Advanced Solid Tumors; Breast Cancer; Inflammatory Breast Cancer; Castleman's Disease; Multiple Myeloma
Keywords: Inflammatory breast cancer; Castleman's Disease; Multiple Myeloma; Breast cancer; Solid tumors; CK2 inhibitor
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms; Castleman Disease; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CX-4945 oral formulation — CX-4945 Capsules, Oral, Dose escalation study, Dose schedule: twice daily or four times daily for 21 consecutive days every 28 days.

SUMMARY:
This Phase 1 study of oral CX-4945 is designed to test the safety, tolerability and highest safe dose level of this CK2 inhibitor in patients with advanced solid tumor cancers, Castleman's Disease or Multiple Myeloma.

DETAILED DESCRIPTION:
Elevated CK2 activity has been associated with malignant transformation and aggressive tumor growth and overexpression of CK2 has been documented in multiple types of cancer. CK2 has emerged as a potential anticancer target and inhibition of CK2 represents a potential therapeutic strategy to target a specific molecular defect perpetuating many cancers. CX-4945 has demonstrated potent inhibition of CK2 enzymatic activity. This study will evaluate the safety, pharmacokinetics (PK), and pharmacodynamic (PD) effects of CX-4945 administered to patients with malignancies or lymphoproliferative disorders known to overexpress CK2 including advanced solid tumors, Multiple Myeloma and Castleman's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignancy or lymphoproliferative disorder known to over express CK2 which has failed standard therapies (surgery, radiotherapy, endocrine therapy, chemotherapy) or for which effective therapy is not available, including the following types: (examples)

  * Lung cancer
  * Renal cell cancer
  * Breast cancer
  * Inflammatory breast cancer
  * Head and neck cancer - squamous cell
  * Prostate cancer
  * Colorectal cancer
  * Castleman's disease (multi-centric disease)
  * Multiple myeloma (Eligible patients must have quantifiable M-protein levels present in serum and/or urine)
* At least 18 years of age.
* One or more tumors measurable on radiograph or CT scan, or evaluable disease defined as non-measurable lesions per RECIST or detection of protein M in serum and/or urine of patients with Multiple Myeloma (serum ≥ 10 gm/L and urine ≥ 200 mg/24 hr).
* Laboratory data as specified below:
* Hematology: ANC >1500 cells/mm3, platelet count >100,000 cells/mm3 and Hemoglobin > 9 gm/L
* Hepatic: bilirubin <1.5 X ULN; alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 2.5 X ULN. Patients with known liver metastases or liver neoplasms: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 5.0 X ULN
* Renal: serum creatinine within normal limits (WNL), defined as within 10% of the institution's stated reference range, or a calculated creatinine clearance >60 mL/min/1.73 m2 for patients with abnormal, increased, creatinine levels. Patients with Multiple Myeloma (only): serum creatinine ≤ 2.5 the institutional upper limit of the normal range and a calculated creatinine clearance > 40 mL/min/1.73 m2.
* Coagulation: INR < 1.5 times normal, aPTT < 1.5 times normal. Patients receiving therapeutic doses of anticoagulant therapy may be considered eligible for the trial if INR and aPTT are within the acceptable therapeutic limits for the institution.
* A negative pregnancy test (if female of childbearing potential).
* Estimated life expectancy of at least 3 months
* Karnofsky Performance Status ≥ 70%
* For men and women of child-producing potential, use of effective contraceptive methods during the study
* Ability to understand the requirements of the study, provide written informed consent.

Exclusion Criteria:

* Pregnant or nursing women.
* Seizure disorders requiring anticonvulsant therapy.
* Known brain metastases (unless previously treated and well controlled for a period of > or = 3 months).
* Major surgery, other than diagnostic surgery, within 4 weeks prior to the first dose of test drug.
* Treatment with radiation therapy or surgery within one month prior to study entry
* Treatment with chemotherapy or investigational drugs within 21 days prior to the screening visit. Acute toxicities from prior therapy must have resolved to Grade ≤ 1 above baseline.
* Patients with a history of a second malignancy within 3 years of the baseline visit excluding cutaneous carcinomas and in-situ carcinoma.
* Concurrent severe or uncontrolled medical disease.
* Active symptomatic fungal, bacterial and/or viral infection including active HIV or viral hepatitis.
* Difficulty with swallowing or an active malabsorption syndrome
* Chronic diarrhea
* Gastrointestinal diseases including gastritis, ulcerative colitis, Crohn's disease, or hemorrhagic coloproctitis
* History of gastric or small bowel surgery involving any extent of gastric or small bowel resection.
* Clinically significant bleeding event within the last 3 months, unrelated to trauma, or underlying condition that would be expected to result in a bleeding diathesis
* Patients who have exhibited allergic reactions to a similar structural compound or to a formulation component.
* Concomitant use of warfarin and HMG-CoA reductase inhibitors (statins)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Safety (Dose limiting toxicities, maximum tolerated dose) | One year (Assessed at Cycle 1)
Drug-related adverse events | One Year (Asessed from first administration of study drug through 30 days after the last dose)

SECONDARY OUTCOMES:
Pharmacokinetic and pharmacodynamic assessments | One Year (Assessed during Cycle 1)
Observe evidence of antitumor activity | One Year (Assessed after every two cycles)
Establish the recommended Phase 2 dose | One Year (Study completion)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Cylene Pharmaceuticals
Locations (4):
- United States (4):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Front Range Cancer Specialists, Loveland, Colorado
  - U T M D Anderson Cancer Center, Houston, Texas